CLINICAL TRIAL: NCT05222165
Title: A Phase 1b/2, Multicenter, Open-Label Study of Oral Infigratinib in Pediatric Subjects With Advanced Solid and Central Nervous System (CNS) Tumors (Phase 1b) and in Subjects With Recurrent or Progressive Low-Grade Gliomas Harboring Selected FGFR1, FGFR2, or FGFR3 Alterations (Phase 2)
Brief Title: Study With Infigratinib in Subjects With Advanced Solid and CNS Tumors or Recurrent or Progressive Low-Grade Glioma With Selected FGFR1-3 Alterations
Acronym: NEWEL
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The company decided to interrupt the development of the drug in all oncological indications
Sponsor: Helsinn Healthcare SA (Industry)
Collaborators: Labcorp Corporation of America Holdings, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INFI-21-07; 2021-005614-34 (EudraCT Number)
Record Dates: First submitted 2022-01-12; First posted 2022-02-03 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Advanced Solid Tumor; CNS Tumor; Recurrent WHO Grade II Glioma
Keywords: Low-Grade Glioma; FGFR1-3 Mutation or fusion/rearrangements; FGFR1-3 Fusion; FGFR1-3 Rearrangements; Advanced Solid Tumor; CNS Tumor
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — infigratinib

STUDY DESIGN:
Intervention Model Description: Phase 1b: Rolling 6 design, 3 cohorts Phase 2: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Infigratinib (BGJ398) (Experimental): Generic name: infigratinib. Dosage forms: 18mg and 25mg sprinkle capsules and 25mg, 75mg, 100mg capsules.
  Phase 1b Three dose levels escalation until RP2D is determined.
  Phase 2
  * Pediatric patients: dose defined in the phase 1b (RP2D);
  * Adults: 125 mg.
  Frequency: once daily for 21 days in each 28-day treatment cycle.
  Duration: Treatment duration will last up to 26 cycles unless progression, death or unacceptable toxicity occur.
  Interventions: Drug: Infigratinib

INTERVENTIONS:
Drug: Infigratinib — Hard gelatin capsules for oral use
  Other Names: BGJ398

SUMMARY:
The phase 1b study is aimed at determining the pediatric recommended phase 2 dose (RP2D) of Infigratinib.

The phase 2 study will evaluate efficacy and safety of infigratinib.

DETAILED DESCRIPTION:
Phase 1b:

Pediatric subjects with advanced solid and CNS tumors or recurrent or progressive Low-Grade Glioma with selected FGFR1-3 alterations will follow a standard dose escalation, in 3 dose levels, to determine the pediatric recommended Phase 2 dose (RP2D) and to assess the safety.

Dose escalation decisions will be assessed through three dose level cohorts.

Phase 2:

To evaluate the efficacy and safety in Pediatric and adult subjects with LGG with selected FGFR1-3 alterations (including subjects who received infigratinib at the RP2D).

ELIGIBILITY:
Inclusion Criteria:

Phase 1b:

* Subject must be ≥ 3 to <18 years of age at the Screening visit.
* Confirmed diagnosis of one of the following:

  1. LGG (WHO Grade I or II glioma) based on histology, molecular, and clinical criteria concordant with the WHO Grading of Tumors of the Central Nervous System, including glial or mixed neuronal-glial tumor
  2. Histologically/cytologically confirmed CNS tumor (other than LGG).
  3. Histologically/cytologically confirmed advanced solid tumor.
* Disease is recurrent or progressive after standard therapy (at least 1 prior standard therapy appropriate for tumor type and stage of disease unless available standard therapies are considered inadequate for the subject).

Phase 2 at screening:

* Diagnosis of recurrent or progressive (at least 1 prior standard therapy) LGG (WHO Grade I or II glioma), including glial or mixed neuronal-glial tumor, based on histology, molecular, and clinical criteria concordant with the WHO Grading of Tumors of the Central Nervous System.
* Age 3 years and older at screening visit.

Phase 1b/2 (all subjects) at screening:

* Able to swallow and retain oral medication.
* Willing to stop consumption of grapefruit, grapefruit juice, grapefruit hybrids, pomegranates, star fruits, pomelos, Seville oranges, or products containing juice of these fruits; and have not consumed these within 7 days before the first dose of study drug.
* Willing and able to comply with scheduled visits, treatment plan, and laboratory tests.

Sex and Contraceptive/Barrier Requirements

* Contraceptive and barrier use as well as pregnancy testing is required as appropriate for the age and sexual activity of pediatric and adult subjects and as required by local regulations.
* Subjects can be male and female.
* A legal guardian or caregiver must be able to accurately maintain the pediatric subject's take-home record, including items of general health.

Exclusion Criteria:

* Prior treatment with a FGFR1-3 selective inhibitor.
* Known serious active infection or any clinically significant systemic illness, which in the Investigator's opinion, cannot be adequately controlled with appropriate therapy or would compromise the subject's ability to tolerate the study drug.
* Received anti-convulsant drugs that are strong inducers of CYP3A4 (i.e., carbamazepine, phenobarbital, phenytoin) within 4 weeks before starting study treatment.
* Currently receiving treatment with agents that are known strong and moderate inducers of CYP3A4 within 4 weeks from start of treatment or inhibitors of CYP3A4 within 1 week from start of treatment, including herbal preparations; medications which increase serum phosphorus and/or calcium concentration; use of a proton-pump inhibitors (e.g., omeprazole) within 4 days prior to start of study therapy or H2 receptor antagonists (e.g., famotidine) within 2 days prior to the start of study therapy.
* Uncontrollable seizures.
* Have current evidence of corneal or retinal disorder/keratopathy including, but not limited to, bullous/band keratopathy; corneal abrasion, inflammation, or ulceration; or keratoconjunctivitis, confirmed by ophthalmic examination. Subjects with asymptomatic ophthalmic conditions assessed by the Investigator to pose minimal risk for study participation may be enrolled in the study.
* Have current evidence of endocrine alterations of calcium/phosphate homeostasis (e.g., parathyroid disorders, history of parathyroidectomy, tumor lysis, tumoral calcinosis), unless well controlled.
* Have a history and/or current evidence of extensive tissue calcification including, but not limited to, the soft tissue, kidneys, intestine, vasculature, myocardium, and lung with the exception of calcified lymph nodes, minor pulmonary parenchymal calcifications, small renal cyst or stone calcifications, and asymptomatic coronary calcification.
* Have impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral infigratinib (e.g., active ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection).
* Had major surgery within 2 weeks of enrollment or not fully healed from open wound.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Phase 1b Dose Limiting Toxicity (DLT) rate | 28 days
  An adverse event (AE) or abnormal laboratory value that are not clearly due to the underlying disease or extraneous causes, including those AEs and abnormal laboratory values that result in a failure to meet the criteria for re-treatment.
Phase 2 Objective Response Rate (ORR) by Blinded Independent Central Review (BICR) | Up to 24 months
  The proportion of subjects who achieve a confirmed complete response (CR), confirmed partial response (PR), or confirmed minor response (MR) for subjects with LGG. For other subjects, ORR is defined as proportion of subjects who achieve a confirmed CR or confirmed PR.

SECONDARY OUTCOMES:
Phase 1b Pharmacokinetics (PK): Cmax | Up to 24 months
  The maximum observed plasma concentration after drug administration (defined as the 2-hour post-dose concentration)
Phase 1b Pharmacokinetics (PK): AUC | Up to 24 months
  Area under the plasma concentration-time curve
Phase 1b Pharmacokinetics (PK): T1/2 | Up to 24 months
  Apparent terminal Half-Life
Phase 1b Pharmacokinetics (PK): Tmax | Up to 24 months
  Peak time
Phase 1b Pharmacokinetics (PK): CL/F | Up to 24 months
  Apparent clearance Day1
Phase 1b Pharmacokinetics (PK): Vz/F | Up to 24 months
  Apparent volume of distribution
Phase 1b Best Overall Response (BOR) assessed by Investigator | Up to 24 months
  The best response recorded from the start of the study treatment until the end of treatment taking into account any requirement for confirmation.
Phase 1b Disease Control Rate (DCR) assessed by Investigator | Up to 24 months
  The proportion of subjects with a Best Overall Response (BOR) of complete response (CR), partial response (PR), minor response (MR) or standard deviation (SD) for subjects with LGG. For other subjects, DCR is defined as the proportion of subjects with a BOR of CR, PR or SD.
Phase 1b Objective Response Rate (ORR) assessed by Investigator | Up to 24 months
Phase 1b Duration of Response (DOR) assessed by Investigator | Up to 24 months
  The time from first documentation of objective response (partial response (PR), complete response (CR), minor response (MR)) to first documentation of PD or death due to any cause, whichever occurs first.
Phase 1b Time to Response (TTR) assessed by Investigator | Up to 24 months
  The time from the date of the start of the treatment to the date of the first documented objective response (partial response (PR), complete response (CR), minor response (MR)) which is subsequently confirmed.
Phase 1b Progression Free Survival (PFS) assessed by Investigator | Up to 24 months
  The time from the date of the start of treatment to the date of the first documented progression or death due to any cause, whichever is earlier.
Post-treatment termination Phase 1b Progression Free Survival (PFS) assessed by Investigator | After treatment termination up to progression disease (PD), assessed for further 24 months
  PFS after treatment termination is the time from the date of treatment interruption for any reason excluding progression disease (PD) to the date of the first documented progression or death due to any cause, whichever is earlier.
Phase 1b Best change in tumor size assessed by Investigator | Up to 24 months
  The minimum change from baseline in the sum of diameters of target lesions.
Phase 2 Duration of Response (DOR) assessed by blinded independent central review (BICR) | Up to 24 months
Phase 2 Time to Response (TTR) assessed by blinded independent central review (BICR) | Up to 24 months
Phase 2 Progression Free survival (PFS) assessed by blinded independent central review (BICR) | 6 months from treatment initiation
Phase 2 Progression Free survival (PFS) assessed by blinded independent central review (BICR) | 12 months from treatment initiation
Phase 2 Progression Free survival (PFS) assessed by blinded independent central review (BICR) | 24 months from treatment initiation
Post-treatment termination Phase 2 Progression Free survival (PFS) assessed by blinded independent central review (BICR) | After treatment termination up to progression disease (PD), assessed for further 24 months
Phase 2 Overall Survival (OS) | 12 months
  Overall Survival (OS) is defined as the time from the date of start of treatment to the date of death due to any cause.
Phase 2 Overall Survival (OS) | 24 months
Phase 2 Best Overall Response (BOR) assessed by blinded independent central review (BICR) | Up to 24 months
Phase 2 Disease Control Rate (DCR) assessed by blinded independent central review (BICR) | Up to 24 months
Phase 2 Best change in tumor size assessed by blinded independent central review (BICR) | Up to 24 months
Phase 2 Best Overall Response (BOR) assessed by Investigator | Up to 24 months
Phase 2 Disease Control Rate (DCR) assessed by Investigator | Up to 24 months
Phase 2 Objective Response Rate (ORR) assessed by Investigator | Up to 24 months
Phase 2 Duration of Response (DOR) assessed by Investigator | Up to 24 months
Phase 2 Time to Response (TTR) assessed by Investigator | Up to 24 months
Phase 2 Progression Free Survival (PFS) assessed by Investigator | Up to 24 months
Phase 2 Best change in tumor size assessed by Investigator | Up to 24 months
Post-treatment termination Phase 2 Progression Free Survival (PFS) assessed by Investigator | After treatment termination up to progression disease (PD), assessed for further 24 months
Phase 1b Incidence/severity of Adverse Events (AEs) | Up to 30 days after treatment termination
  Number of patients who experienced AEs to assess the safety and tolerability of infigratinib in subjects with recurrent or progressive LGG.
Phase 2 Incidence/severity of Adverse Events (AEs) | Up to 30 days after treatment termination
Phase 1b Incidence/severity of Serious Adverse Events (SAEs) | Up to 30 days after treatment termination
  Number of patients who experienced SAEs to assess the safety and tolerability of infigratinib in subjects with recurrent or progressive LGG.
Phase 2 Incidence/severity of Serious Adverse Events (SAEs) | Up to 30 days after treatment termination

CONTACTS AND LOCATIONS:
Locations (10):
- United States (6):
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - Children's National Hospital - Brain Tumor Institute, Washington D.C., District of Columbia
  - Nicklaus Children's Hospital, Miami, Florida
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke Cancer Institute (DCI) - The Preston Robert Tisch Brain Tumor Center, Durham, North Carolina
  - UPCM - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
- Canada (3):
  - University of Alberta - Stollery Children's Hospital (SCH), Edmonton, Alberta
  - McMaster Children's Hospital (MCH), Hamilton, Ontario
  - University of Toronto - The Hospital for Sick Children (SickKids), Toronto, Ontario
- Universitaetsklinikum Heidelberg (UKHD) - Zentrum fuer Kinder- und Jugendmedizin - Klinik Kinderheilkunde III, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No